CLINICAL TRIAL: NCT05170880
Title: Effect of Primary Non-surgical Endodontic Therapy on Glycaemic Control in Type 2 Diabetic Patients With Asymptomatic Apical Periodontitis: A Randomized Controlled Trial
Brief Title: Effect of Primary Non-surgical Endodontic Therapy on Glycaemic Control in Type 2 Diabetic Patients With Asymptomatic Apical Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Dr. Aparna
Record Dates: First submitted 2021-12-11; First posted 2021-12-28 (Actual); Last update posted 2021-12-28 (Actual); Status verified 2019-01

CONDITIONS: Diabete Type 2; Apical Periodontitis
Keywords: Type 2 Diabetes Mellitus, Apical Periodontitis
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Periapical Periodontitis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): After fulfilling the eligibility criteria, patients will be informed about the study and written consent to participate in the study will be acquired from each patient after explaining risks, benefits and alternative treatments.The endodontic treatment for all patients will be performed by a single operator (S.A) following a standardized protocol.
  Interventions: Procedure: Primary endodontic treatment
- Control Group (No Intervention): The control group will receive no endodontic treatment during the study period. After completion of the study, these patients will be given primary non-surgical endodontic treatment.

INTERVENTIONS:
Procedure: Primary endodontic treatment — Primary non surgical endodontic treatment will be provided to patients in treatment group.
  Arms: Treatment Group

SUMMARY:
To evaluate the effect of primary non-surgical endodontic therapy on glycaemic control in type 2 diabetic patients with asymptomatic apical periodontitis.After fulfilling the eligibility criteria, patients will be informed about the study and written consent to participate in the study will be acquired from each patient after explaining risks, benefits and alternative treatments.The endodontic treatment for all patients will be performed by a single operator (S.A) following a standardized protocol. The control group will receive no endodontic treatment during the study period. After completion of the study, these patients will be given primary non-surgical endodontic treatment. The patients in control group will be rendered the necessary treatment, if they become symptomatic and/or deny the consent during the course of the study. These patients will be excluded from the study.

DETAILED DESCRIPTION:
INTRODUCTION:

Diabetes mellitus (DM) is a clinically and genetically heterogeneous group of disorders affecting the metabolism of carbohydrate, lipid or proteins, in which hyperglycemia is the main feature. These disorders are either due to insulin deficiency related to autoimmune destruction of pancreatic beta cells (type 1) or target tissue resistance to its cellular metabolic effects (type 2).1 Patients suffering from DM are known to have increased susceptibility to infections2.Evidence has consistently indicated that DM is a risk factor for increased severity of periodontal disease3,4.

Apical Periodontitis (AP) is an acute or chronic inflammation of the periodontium located at the root apex caused by bacterial infection of the pulp canal system5.

Traditionally, DM is diagnosed by either fasting or postprandial blood glucose but since 2010 American Diabetes Association (ADA) has recommended mean HbA1c as diagnostic criteria of diabetes with its threshold level of 6.5%. HbA1c is a resulting product of hemoglobin and glucose interaction and its elevated level indirectly reflects the hyperglycemic condition i.e. DM. Studies have been conducted linking periodontal disease and diabetes mellitus in terms of prevalence and worsening of glycemic control in diabetics as well as effect of periodontal treatment on glycemic control in diabetic patients. Nevarro-Sanchez et al showed significant improvement in HbA1c levels after non surgical periodontal therapy in diabetic patients .

The aim of the present trial is to evaluate the effect of endodontic therapy on glycemic status in patients with apical periodontitis.

AIM AND OBJECTIVES:

To evaluate the effect of primary non-surgical endodontic therapy on glycaemic control in type 2 diabetic patients with asymptomatic apical periodontitis.

MATERIALS AND METHODOLOGY:

This study will be conducted in the department of conservative dentistry and endodontics, Post Graduate Institute of Dental Sciences (PGIDS), Rohtak. Study subjects will be obtained from the pool of OPD patients in the Department of conservative dentistry and endodontics, PGIDS, Rohtak.

Study Design: Intervention Study period: December Study subjects: 30

Baseline parameters -- Endodontic evaluation - Pulp sensibility testing will be performed with a combination of heat test, cold test and electric pulp test. Teeth not responding to both thermal and electric test will be considered non vital.

Radiographic evaluation - Radiographs with paralleling cone technique at baseline and at subsequent appointment (3 months) will be taken at standardized exposure parameters.

Glycemic Control Assessment To determine the metabolic control status of diabetic patients, HbA1c will be registered on the day of treatment initiation. For the metabolic assessment, venous blood samples will be taken from each patient and analysed for glycated haemoglobin (HbA1c). Metabolic measurements will be performed at baseline and at 3rd month following the endodontic treatment in the treatment and control group.

Randomization: Patients will be randomly allocated by envelope method into two groups- intervention group (IG) , Group II= Control group (CG). The opaque envelopes will be prepared by an independent observer blinded to the treatment groups. The patients will be asked to choose an envelope at the time of recruitment which will decide the group into which patient will be allocated.

Methodology:

After fulfilling the eligibility criteria, patients will be informed about the study and written consent to participate in the study will be acquired from each patient after explaining risks, benefits and alternative treatments. Prior to treatment a thorough clinical and radiological examination will be carried out and thorough history will be taken from each patient. Patients will be instructed to continue with their medical treatment of DM (oral hypoglycemic agents), diet and life style without modifications during the study period.

Clinical Procedure:

The endodontic treatment for all patients will be performed by a single operator (S.A) following a standardized protocol. After local anesthesia administration (2 % xylocaine with 1:80000 epinephrine), access cavity will be prepared using under rubber dam isolation. After pulp chamber debridement and canal orifices identification, coronal shaping & enlargement will be performed with low speed gates-glidden drills to obtain straight line access to the apical third of each root canal. Working length will be determined with the help of Root ZX apex locator and verified radiographically. Canals will be prepared using the crown down technique with rotary instruments. Canals will be irrigated with 5 ml of 5.25 % sodium hypochlorite (NaOCl) subsequent to change of each instrument. After complete canal instrumentation, the canals will be irrigated with 5.0 ml of 17% ethylene-diaminetetra acetic acid for 1 minute followed by a final irrigation with 5.0 ml of 5.25% NaOCl. Canals will be filled with a paste of calcium hydroxide and access will be sealed temporarily with Intermediate Restorative Material. Patient will be scheduled for second visit after one week. At the next appointment, the paste will be removed with Hedstrom files followed by copious irrigation with 5.25% NaOCl. Canals will be obturated using lateral condensation technique. After obturation, the cavity will be permanently restored. Immediate post-operative radiograph will be taken using preset exposure parameters with a Rinn paralleling device.

The control group will receive no endodontic treatment during the study period. After completion of the study, these patients will be given primary non-surgical endodontic treatment. The patients in control group will be rendered the necessary treatment, if they become symptomatic and/or deny the consent during the course of the study. These patients will be excluded from the study.

Post - Operative Follow-Up:

Patients will be evaluated after 3 months. Radiograhic evaluation: periapical radiographs will be taken to observe the healing.

Metabolic evaluation: For the metabolic assessment patients will be analysed for glycated haemoglobin (HbA1c).

Clinical evaluation: Patients will be evaluated for the presence of any abnormal clinical findings.

Statistical analysis Shapiro Wilk test will be used to analyze the distribution of data. Categorical data will be analyzed by chi square test. Regression analysis will be done to observe any association between independent and dependent variables. Interobserver/intraobserver reliability will be analyzed with Cohen kappa analysis

ELIGIBILITY:
Inclusion Criteria:

Patient willing to participate in the study. Patients with a history of type 2 DM (with HbA1c ≥ 6.5%), between the age of 30 to 65 years, asymptomatic mature permanent teeth with pulpal necrosis as confirmed by a negative response to cold and electric test and radiographic evidence of AP no history of systemic antibiotic administration within the last 1 month;

Exclusion Criteria:

Symptomatic patients Retreatment Unwillingness of patients Procedural errors and calcified canals ,inability to achieve apical patency in any canals Immuno-compromised, pt. on long term steroids, pregnant and patient with any other systemic illness except diabetes mellitus.

Teeth with periodontal disease.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-02-11 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
HbA1c levels | 3 months
  Glycemic status will be evaluated using HbA1c levels.

CONTACTS AND LOCATIONS:
Locations (1):
- Post Graduate Institute of Dental Sciences, Rohtak, Haryana, India

IPD SHARING:
Plan to Share IPD: No